CLINICAL TRIAL: NCT00569881
Title: Effect of Gatifloxacin 0.3% and Moxifloxacin 0.5% on Epithelial Wound Healing After Photorefractive Keratectomy
Brief Title: Effect of Topical Fluoroquinolones on Epithelial Wound Healing After PRK
Status: Completed | Type: Observational
Sponsor: Donnenfeld, Eric, M.D. (Individual)
Responsible Party: Eric Donnenfeld, MD, Founding Partner, OCLI
Other Study IDs: Donnenfeld2
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Corneal Epithelial Wound Healing
Keywords: Epithelium; Wound Healing; PRK
MeSH Terms: interventions — Gatifloxacin; Moxifloxacin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Corneal epithelial wound healing with moxifloxacin
  Interventions: Drug: gatifloxacin and moxifloxacin
- 2: Corneal epithelial wound healing with gatifloxacin
  Interventions: Drug: gatifloxacin and moxifloxacin

INTERVENTIONS:
Drug: gatifloxacin and moxifloxacin — Comparison of wound healing between drugs
  Other Names: Zymar and Vigamox

SUMMARY:
The prescribed antibiotic for prophylaxis of infection following PRK should be effective at eradicating a potential infection. In addition, the antibiotic should have a rapid onset of action, effectively penetrate the target tissue, and be safe and not toxic to any layer of the healing cornea, especially the epithelium. Several studies have investigated the toxicity of the fourth generation fluoroquinolones on the corneal epithelium and studies have demonstrated that gatifloxacin is less deleterious to the healing cornea than moxifloxacin. Most of these studies, however, have been conducted in animals. This was a retrospective chart review.

DETAILED DESCRIPTION:
Prior generation fluoroquinolones predominantly either inhibit topoisomerase II (DNA Gyrase) or topoisomerase IV and therefore only require one genetic mutation for bacteria to develop resistance. Fourth-generation fluoroquinolones are equally effective against topoisomerase II and IV, which significantly expands their spectrum of action against gram-positive agents and atypical mycobacteria and Nocardia . This duality of action of the fourth generation fluoroquinolones requires that for bacteria to become resistant to these agents, the bacteria must undergo two genetic mutations resulting in a significantly decreased chance of an organism developing resistance.Minimum inhibitory concentrations determined in vitro suggest that fourth-generation fluoroquinolones are more effective than second- and third-generation fluoroquinolones against gram-positive bacteria including Staphylococcal species found in endophthalmitis and bacterial keratitis cultures. The increased efficacy of fourth-generation fluoroquinolones make these antibiotics important agents to evaluate for prophylaxis against post-PRK infections. This was a retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for inclusion if they were a healthy male or female 18 years of age or older and were candidates for bilateral PRK.
* Eligible patients had a best-corrected Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity score equivalent to a Snellen score of 20/30 or better in each eye, had a stable prescription for 1 year, were willing to participate in the study, and were able to comprehend and sign the informed consent form.
* All subjects were instructed that if they decide not to participate they could withdraw from the study at any time.

Exclusion Criteria:

* Patients were excluded from the study if they had a history of refractive or other ocular surgery in either eye.
* Patients with any condition which could delay wound healing were not eligible to participate.
* They were excluded if they had poor tolerance to any component of the masked study fluoroquinolones, Acular® LS (Allergan) or Pred Forte® (Allergan).
* Patients were also excluded if they required the use of a systemic antibiotic during the study period, were involved in another investigational study or had participated in a study within 30 days prior to the start of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presented to the practice of a cornea trained ophthalmic consultant.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2007-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Wound Healing | Days after PRK

CONTACTS AND LOCATIONS:
Overall Officials: Eric Donnenfeld, MD, Principal Investigator — OCLI